CLINICAL TRIAL: NCT03786835
Title: Healthy Older People Everyday (HOPE) - Role of Healthy Diet on Muscle and Bone Health
Acronym: HOPE-DIET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Health Promotion Board (HPB) (Unknown); Saw Swee Hock Shool of Public Health, National University of Singapore (Unknown)
Responsible Party: Principal Investigator, Medicine, Head & Senior Consultant, Division of Geriatric Medicine, National University Hospital, Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/01183
Record Dates: First submitted 2018-12-11; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Muscle Weakness; Bone Health; Cognitive Decline
MeSH Terms: conditions — Muscle Weakness; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No intervention) (No Intervention): Participants will not undergo any treatment. Continue with usual daily activities and diet for 6 months.
- Nutrition group (Experimental): Participants will receive protein enriched food to supplement the diet for 6 months.
  Interventions: Other: Protein supplementation and regular physical activity
- Exercise group (Experimental): Participants will exercise 3 times a week for 60 minutes each time over 6 months.
  Interventions: Other: Protein supplementation and regular physical activity
- Nutrition + Exercise group (Experimental): Participants will receive protein enriched food to supplement the diet and exercise 3 times a week for 60 minutes each time over 6 months.
  Interventions: Other: Protein supplementation and regular physical activity

INTERVENTIONS:
Other: Protein supplementation and regular physical activity — To determine if high protein diet and/or regular physical activity improves muscle and bone health
  Arms: Exercise group; Nutrition + Exercise group; Nutrition group

SUMMARY:
Certain clinical syndromes eg frailty, sarcopenia, dementia, depression, cognitive impairment, vision impairment and falls in older adults carry an increased risk for poor health outcomes and if identified early, can be prevented, delayed or reversible. There is evidence to suggest that exercise and dietary intervention can help delay or prevent sarcopenia, frailty and dementia.

The current hypothesis is older adults do not consume enough protein in their diet. Local delicacies enhanced with protein content, in addition to physical activity will improve muscle strength, function, perceived health status and possibly may even reverse frailty and sarcopenia. Additionally, it is hypothesized that combination of multi component group exercise activities and high protein nutrition will be effective in improving participants' social, mental and physical status.

DETAILED DESCRIPTION:
From our own published local data, the prevalence of pre-frailty in North-West area is 37% and frailty 6.2%. Prevalence of frailty in individuals with diabetes is 12%, double that of general population.

Evidence suggest that multi-component intervention may delay the onset of disability, and in some cases reverse frailty with the potential to avert preventable adverse events such as falls, fractures and reduce overall healthcare utilisation and extend health-span. There is a similar multi-centre trial in progress in Europe called SPRINTT. As physical exercise and adequate protein and energy intake are to date the only strategies of proven efficacy to improve muscle health, it is important that we develop locally relevant protein enriched food prototypes that can deliver an effective dosage of protein to the older adult and compare them with available protein enriched supplements. High protein diet stimulates muscle protein synthesis and plays a role in delaying the onset of frailty and sarcopenia. An adequate intake of dietary proteins is vital to maintaining muscle mass and stimulating protein synthesis. Older adults are at high risk for insufficient protein intake and furthermore, the current recommended dietary allowance for protein (0.8 g/kg/day) might not be sufficient for preserving muscle mass and quality in old age. It appears therefore appropriate to promote a protein intake of 1.0-1.2 g/kg/day, while 1.2-1.5 g/kg/day of protein may be required in older adults with acute or chronic diseases. Finally, older people with severe illnesses or overt malnutrition may need as much as 2.0 g/kg/day of protein. In addition to protein, the PROVIDE study also showed that sufficient levels of vitamin D and protein is necessary to increase muscle mass and reduce sarcopenia. While most middle aged adults and older adults attempt to keep up with physical activity, very few actually are aware of importance of protein and Vitamin D enriched diet. Exercise and increased protein intake can also down-regulate systemic inflammation.

Locally, there's one small study (n=49 for nutrition and n=49 combined intervention) which documented reversal of frailty with multicomponent intervention, where the nutrition component was a commercial formula Fortisip (Nutricia Dublin). Up to now, there are no locally developed high protein supplements and we have no data on average protein content of local diet consumption in older adults. If locally produced, culturally-relevant high protein food prototype is widely accepted and is proven to improve function and quality of life, it will be an innovative solution to solving nutritional gaps and delivering an effective dose of protein to the elderly population in Singapore. This can especially help the elderly population receive protein supplementation not through commercially produced expensive supplements but through the foods and drinks that they consume everyday. These prototypes can also help the local food and beverage industry recognize the importance and value of investing resources into the continued development of these products to better address local public health needs and possibly export these products to the wider region's ageing population.

In addition, the results from this study will provide the basis and baseline for a review of the current recommended dietary allowance for protein, especially among older adults. The current recommendation of 0.8 g of protein/kg/day was based on the maintenance of a healthy adult's nitrogen balance. It would be important to formulate a set of recommendation to meet the functional and physiological needs of the elderly.

This programme will be the nutritional arm of a current study called 'HAPPY' Healthy Ageing Promotion Program For You, where participants are screened for frailty in the day care, senior activity centre's and community centre's. Participants with cognitive impairment and / or pre-frail are invited to participate in dual task exercise led by trainer from Japan. This locally produced high protein food will be trialled in these participants who have been identified during screening for "HAPPY". Informed consent will be obtained from participants to participate in the HAPPY and HOPE programmes.

ELIGIBILITY:
Inclusion Criteria:

* At least pre-frail (Frail scale score of at least 1) but ambulant
* Grip strength not more than 25kg for males and 18kg for females

Exclusion Criteria:

* With kidney conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in frailty status | 2 years
  Changes in frailty status by 5-item FRAIL scale Scale range from 0 to 5, the higher the value, the more frail.
Changes in lower extremity physical performance | 2 years
  Changes in short physical performance battery (SPPB) summary score 3 subscales (range from 0 to 4 for balance, gait speed and chair stand) summed to give total score range from 0 to 12.
  The higher the value, the better the performance of lower extremity.

SECONDARY OUTCOMES:
Changes in upper extremity muscle strength | 2 years
  Changes in handgrip strength test performance (kg)
Changes in skeletal muscle mass | 2 years
  Changes in skeletal muscle mass by bioelectrical impedance analysis
Changes in sarcopenic status | 2 years
  Changes in sarcopenic status by SARC-F scale Scale range from 0 to 10, the higher the value, the greater the likelihood of sarcopenic
Changes in mood | 2 years
  Changes in Geriatric Depression Scale (GDS) Scale range from 0 to 15, the higher the score, the greater the likelihood of depression.
Changes in mood | 2 years
  Changes in UCLA Loneliness Scale Scale range from 0 to 9, the higher the value, the greater the loneliness Scale from 0 to
Changes in cognitive function | 2 years
  Changes in Mini Mental State Examination (MMSE) score 5 subscales: Orientation (0 to 10), Registration (0 to 3), Attention and Calculation (0 to 5), Recall (0 to 3), Language and Praxis (0 to 9) Total scale range from 0 to 30, the higher the value, the less cognitive impairment.
Changes in cognitive function | 2 years
  Changes in Montreal Cognitive Assessment (MoCA)
Changes in nutritional status | 2 years
  Changes in Mini Nutritional Assessment (MNA) score 2 Subscales: Screening (0 to 14) and Assessment (0 to 16) Total scale range from 0 to 30, the higher the value, the more well nourished.
Changes in functional status (instrumental activities of daily living) | 2 years
  Changes in Instrumental Activities of Daily Living (IADL) score Scale range from 0 to 8, the higher the value, the greater the ability.
Changes in functional status (activities of daily living) | 2 years
  Changes in Activities of Daily Living (ADL) score Scale range from 0 to 6, the higher the value, the greater the ability.
Changes in fall risk | 2 years
  Changes in fall efficacy questionnaire
Incidence of self-reported falls | 2 years
  Number of falls assessed by questionnaires
Changes in quality of life | 2 years
  Changes in EuroQoL-5D (EQ5D) score 5 subscales (1 to 5): Mobility, self-care, usual activities, pain/discomfort, anxiety/depressed Each subscale assessed individually.
Changes in social engagement | 2 years
  Changes in Lubben Social Network Scale. Scale range from 0 to 30, the higher the value, the greater the social engagement
Changes in systemic inflammation | 2 years
  Changes in Tumour necrosis factor alpha (TNF-a)
Changes in systemic inflammation | 2 years
  Changes in Interleukin-10
Changes in systemic inflammation | 2 years
  Changes in Interleukin-6
Changes in phase angle by bioelectrical impedance analysis | 2 years
  Changes in phase angle by bioelectrical impedance analysis
Changes in protein mass | 2 years
  Changes in protein mass by bioelectrical impedance analysis
Changes in level of bone biomarkers | 2 years
  Changes in level of serum sclerotin
Changes in level of bone biomarkers | 2 years
  Changes in level of serum osteocalcin
Changes in level of bone biomarkers | 2 years
  Changes in level of free Vitamin D
Acceptance of protein enriched food by local seniors | 2 years
  Assessed by taste test questionnaire
Cost-effectiveness analysis | 2 years
  Cost effectiveness will be evaluated from the societal perspective. Cost of the program as well as healthcare utilization related to frailty and sarcopenia will be collected. An incremental cost effectiveness ratio will be computed by identifying the additional costs associated with the Intervention Group per additional unit of health outcome (QALYs).

IPD SHARING:
Plan to Share IPD: Undecided